CLINICAL TRIAL: NCT03291353
Title: Phase 0- Pilot Study of Pembrolizumab on Immune Cells in Patient With Refractory Acute Myeloid Leukemia
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: This study has closed due to slow accrual.
Sponsor: Michael Boyiadzis (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Michael Boyiadzis, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-056
Record Dates: First submitted 2017-06-19; First posted 2017-09-25 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AML Patients (Experimental): pembrolizumab 200 mg given IV once every three weeks
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — 200 mg IV given every three weeks
  Other Names: Keytruda

SUMMARY:
This is an open label, single-arm, pilot trial to evaluate the immune effects, safety and tolerability of pembrolizumab in subjects newly diagnosed with acute myeloid leukemia (AML) who have persistent leukemia after induction chemotherapy. Patients must have an ECOG performance status of 0-1. The enrollment target for this study is 10 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on the day of signing informed consent.
3. Patients with newly diagnosed AML based on the World Health Organization classification (21) who have persistent leukemia after a course or more of treatment with induction chemotherapy (the diagnosis of persistent disease, which is defined as >10% blasts by evaluation of bone marrow biopsy or bone marrow aspirate).
4. Left ventricular ejection fraction (LVEF) ≥ 45%
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Demonstrate adequate organ function, all screening labs should be performed within 10 days of treatment initiation.
7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential must be willing to use an adequate method of contraception- Contraception, for the course of the study through 120 days after the last dose of study medication.
9. Male subjects of childbearing potential must agree to use an adequate method of contraception- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Has a diagnosis of Acute Promyelocytic Leukemia (APL) as defined by the World Health Organization
2. Relapsed acute myeloid leukemia
3. Bi-lineage or bi-phenotypic leukemias
4. Prior use of clofarabine or fludarabine
5. Previous allogeneic or autologous hematopoietic cell transplantation or solid organ transplantation
6. Is currently participating in and receiving study therapy, or has participated in a study of an investigational agent and received study therapy, or used an investigational device within 4 weeks of the first dose of treatment.
7. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
8. Has a known history of active TB (Bacillus Tuberculosis)
9. Hypersensitivity to pembrolizumab or any of its excipients.
10. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
11. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
12. Concurrent active malignancy; exceptions include patients who have been disease free for 5 years, patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, or patients with another malignancy that is indolent or definitively treated.
13. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis and/or has known active central nervous system (CNS) leukemia involvement.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
19. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
20. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
21. Has known active Hepatitis B or Hepatitis C.
22. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-08-19 (Estimated); Study Completion 2022-08-19 (Estimated)

PRIMARY OUTCOMES:
Adverse event assessment | From prior to first dose up to 48 months
  Adverse event assessment using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Response Rate (RR) | Up to greater than or equal to 48 months
  The number of patients receiving treatment that experience either a Partial Response (remission) and/or a Complete Response (remission) / the total number of treated patients, per Response Criteria for Acute Leukemia criteria.
Overall survival | Up to greater than or equal to 48 months
  Median overall survival will be estimated by the Kaplan-Meier method with 90% confidence intervals.

OTHER OUTCOMES:
Percent change of neutrophils and lymphocytes | Up to greater than or equal to 48 months
  Percent change of neutrophils and lymphocytes from baseline before therapy to follow up
Absolute number of CD4+ T cells, CD8+ T cells, Treg , NK cells, B cells and monocytes | Up to greater than or equal to 48 months
  Change in number of CD4+ T cells, CD8+ T cells, Treg , NK cells, B cells and monocytes from baseline before therapy to follow up
Absolute number of activated immune effector cells | Up to greater than or equal to 48 months
  Change in number of activated immune effector cells from baseline before therapy to follow up
Levels of TGF-beta and NKG2D ligands | Up to greater than or equal to 48 months
  Change in level from baseline before therapy to follow up

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boyiadzis, MD, MHSc, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States